CLINICAL TRIAL: NCT00849199
Title: Cancer Screening and Prevention Program for High Risk Women
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Lynne Cohen Foundation for Ovarian Cancer Research (Other)
Responsible Party: Sponsor
Other Study IDs: 9541; NYU H#9541 (Other: NYU)
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Ovarian Cancer; Breast Cancer
Keywords: screening; early detection; prevention; cancer; high risk; ovarian cancer; breast cancer
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High risk of breast or ovarian cancer

SUMMARY:
The purpose of this study is to collect information from a large group of women who may have a greater chance to develop cancer because of their own personal history of cancer or because of their family history of cancer.

DETAILED DESCRIPTION:
The objectives of this study are to be a resource of information on women's cancers, including the availability of a genetics counselor for women at risk for hereditary cancer, especially ovarian cancer; to provide referrals for diagnostic tests and appropriate clinics involved in early detection of cancer; to provide access to clinical trials and investigational screening methods in cancer early detection and prevention, whenever applicable; to provide women with educational materials; to develop a database of information compiled from the questionnaires and clinics for use in future studies; to create a registry of family history data from women of diverse racial and ethnic backgrounds who attend our clinic, i.e. who perceive themselves to be at increased risk of breast or gynecologic cancers.Women that participate in the study will be interviewed and asked to fill out a questionnaire. An assessment will then be made based on their information. Based on this assessment, women will be referred to the appropriate clinic or for diagnostic testing or provided with information regarding available protocol studies.

ELIGIBILITY:
Inclusion Criteria:

* Female or male over the age of 18.
* Patients who have a family history of breast and or ovarian cancer.
* Patients who have had a personal history of breast and or ovarian cancer or who themselves or a relative have positive genetic markers for breast or ovarian cancer.
* Patients who seek medical screening and risk assessment for perceived increased risk of breast or ovarian cancer.

Exclusion Criteria:

* Women with psychiatric, psychological or other conditions which prevent fully informed consent.
* Patients seeking medical attention not related to the purposes of this protocol, (e.g. those seeking treatment of a known cancer).
* Women with a history of any medical condition, which places the subject at risk, related to the need for donating blood for research purposes, (e.g., chronic infectious diseases, severe anemia, or hemophilia).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primarily disadvantaged women who have a family history of breast and or ovarian cancer or who have had a personal history of breast and or ovarian cancer or who themselves or a relative have positive genetic markers for breast or ovarian cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1452 (Actual)
Dates: Start 2001-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
To create a registry for women at high risk of breast or ovarian cancer | 15 years

SECONDARY OUTCOMES:
To provide genetic counseling, referrals for diagnostic tests and to appropriate clinics to promote the early detection of cancer; to seek and develop research protocols of early detection and treatment | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Franco Muggia, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Bellevue Hospital, New York, New York
  - NYU Cancer Center, New York, New York
  - NYU Tisch Hospital, New York, New York

REFERENCES:
- [Result] Smith J, Baer L, Blank S, Dilawari A, Carapetyan K, Alvear M, Utate M, Curtin J, Muggia F. A screening and prevention programme serving an ethnically diverse population of women at high risk of developing breast and/or ovarian cancer. Ecancermedicalscience. 2009;3:123. doi: 10.3332/ecancer.2008.123. Epub 2009 Mar 16. PMID 22275995